CLINICAL TRIAL: NCT02121665
Title: Effect of Probiotic Lozenges as an Adjunct to Non Surgical Periodontal Therapy in Chronic Periodontitis Patients: A Randomized Double Blind Placebo Controlled Clinical and Biochemical Study.
Brief Title: Efficacy of a Probiotic Lozenges in Chronic Periodontitis Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CD Pharma India Pvt. Ltd. (Industry)
Collaborators: Government Dental College and Hospital, India (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLOZ/PG/PERIO/2013
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Inersan) Arm (Experimental): Inersan Lozenges (4 Lozenges per day; 1 lozenge in morning,1 lozenge in the afternoon and 2 lozenges in the night). Each probiotic lozenge contains not less than 1 billion CFU of L. brevis CD2
  Interventions: Drug: Probiotic (Inersan)
- Placebo Arm (Placebo Comparator): Placebo Lozenges (4 Lozenges per day; 1 lozenge in morning,1 lozenge in the afternoon and 2 lozenges in the night). Each placebo lozenge contains all excipients except the active constituent (Lactobacillus brevis CD2)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probiotic (Inersan) — Each Inersan lozenge contains not less than 1 billion CFU of Lactobacillus brevis CD2
  Arms: Probiotic (Inersan) Arm
Drug: Placebo — Each placebo lozenge contains all excipients except the active constituent (Lactobacillus brevis CD2)
  Arms: Placebo Arm

SUMMARY:
Periodontal disease is an infectious disease resulting in inflammation within supporting tissues of the teeth, progressive attachment loss, and bone loss. Epidemiological studies reveal that about 10% of the adult population suffer from severe periodontitis.It comprises of two distinct but interconnected etiologic components: the periodontopathic bacteria adjacent to the periodontal tissues, and the host-mediated connective tissue-destructive responses to the causative bacteria and their metabolic products. In the arena of periodontics, the probiotics pose a great potential of plaque modification, halitosis management, altering anaerobic bacteria colonization, improvement of pocket depth, and clinical attachment gain.

Aim of the study is to analyze the beneficial effect of probiotic lozenges as an adjunct to Scaling and Root Planing, on clinical and biochemical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subject of both sexes
* Age group of 25-65 years
* Subjects with generalized moderate to severe chronic periodontitis
* Signed informed Consent

Exclusion Criteria:

* Any known history of systemic diseases
* Patients already on anti-inflammatory drugs or antibiotics
* Patients allergic to any material used in the study
* Pregnant and lactating women
* Periodontal therapy in past 6 months
* Current smoker or smoker in the past

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Improvement in Periodontal Clinical indices | 6 weeks
  Improvement in periodontal clinical indices, namely, Gingival Index (GI), Plaque Index (PI), Probing Pocket Depth (PPD) and Clinical attachment Loss (CAL).

SECONDARY OUTCOMES:
Improvement in biochemical indices | 6 weeks
  Changes in level of inflammatory markers namely PGE2, IL-1beta, TNF-alpha, receptor activator of nuclear factor kappa B ligand (RANKL), Osteoprotegerin (OPG), MMP-9 and MMP-13 in saliva sample

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Sethi, BDS, Principal Investigator — Government Dental College & Hospital, Aurangabad
Locations (1):
- Department of Periodontics, Government Dental College & Hospital, Aurangabad, Maharashtra, India